CLINICAL TRIAL: NCT02881840
Title: An Open Label, Single Dose, Single Period Study to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C] APD421 Administered Via the Intravenous Route to Healthy Male Subjects
Brief Title: Mass-balance Study of [14C]-APD421 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP10020
Record Dates: First submitted 2016-08-01; First posted 2016-08-29 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Post-operative Nausea and Vomiting
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-APD421 (Experimental)
  Interventions: Drug: 14C-APD421

INTERVENTIONS:
Drug: 14C-APD421

SUMMARY:
Open-label, non-randomised, single dose study in 6 healthy male subjects to assess the mass balance recovery, metabolite profile, metabolite identification and pharmacokinetics of 14C-labelled APD421

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 18 to 65 years of age at time of signing informed consent
* Body mass index (BMI) of 18 to 30 kg/m2 or, if outside the range, considered not clinically significant by the investigator
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Must agree to use an adequate method of contraception (as defined in Section 8.4)
* Must have regular bowel movements (ie average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* Prior participation in another study with a radiation burden of > 0.1 mSv and ≤ 1 mSv in the period of 1 year prior to screening; a radiation burden of > 1 mSv and ≤ 2 mSv in the period of 2 years prior to screening; a radiation burden of > 2 mSv and ≤ 3 mSv in the period of 3 years prior to screening, etc (add 1 year per 1 mSv)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Fox, MB BChir, Study Director — Acacia Pharma Ltd
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fox GM, Roffel AF, Hartstra J, Bussian LA, van Marle SP. Metabolism and Excretion of Intravenous, Radio-Labeled Amisulpride in Healthy, Adult Volunteers. Clin Pharmacol. 2019 Dec 2;11:161-169. doi: 10.2147/CPAA.S234256. eCollection 2019. PMID 31819674

RESULTS

PARTICIPANT FLOW:
Groups:
- 14C-APD421: [14C]-APD421 (amisulpride) solution for intravenous infusion (2.5 mg/mL) at 10 mg containing 1.784 MBq (48.2 μCi) 14C administered as a single IV infusion over a 4 minute period.
Period: Overall Study
Arm/Group | 14C-APD421
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 14C-APD421 Amisulpride: Single IV dose administration as an infusion over a 4 minute period
Arm/Group | 14C-APD421 Amisulpride
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: Years]
  Netherlands | 6

OUTCOME MEASURES:

1. Primary Outcome: Mass Balance
Description: Mean recovery of radioactivity in excreta after a single intravenous (IV) dose of carbon-14-labelled APD421
Time Frame: 168 hours
Measure: Mean (Full Range); unit: percent excreted
Arm/Group | 14C-APD421
Number analyzed (Participants) | 6
percent excreted | 96.4 [92.0 to 98.5]

ADVERSE EVENTS:
Time Frame: For the 7 day period after study drug administration
Arm/Group | 14C-APD421
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 14C-APD421 (N=6)
Infusion site pain (General disorders) | 6 (6)
Eye irritation (Ear and labyrinth disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitation or caveats in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No